CLINICAL TRIAL: NCT05309564
Title: Muscle Weakness Duration Post-injection of a Single Dose of Botulinum Toxin in the Masseter Muscle Bilaterally: a One-year Non-randomized Controlled Trial
Brief Title: Muscle Weakness Duration After Single Botulinum Toxin Injection in Masseter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västerbotten (Other Government)
Collaborators: Umeå University (Other); Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTX-Thailand
Record Dates: First submitted 2022-03-14; First posted 2022-04-04 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Bite Force; Botulinum Toxins, Type A
MeSH Terms: interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention with single botulinum neurotoxin injection into masseter.
  Interventions: Drug: Botulinum toxin type A
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Botulinum toxin type A — Single intervention
  Other Names: Xeomin
  Arms: Intervention

SUMMARY:
This study aimed to evaluate the duration of a reduced maximal voluntary bite force after a botulinum toxin intervention. Methods: In an intervention group, 25 units of Xeomin® (Merz Pharma GmbH & Co KGaA, Frankfurt am Main, Germany) botulinum neurotoxin type A were injected into the masseter muscles bilaterally (to a total of 50 units).

DETAILED DESCRIPTION:
This study aimed to evaluate the duration of a reduced maximal voluntary bite force (MVBF) after a botulinum toxin intervention. Methods: In an intervention group, 25 units of Xeomin® (Merz Pharma GmbH & Co KGaA, Frankfurt am Main, Germany) botulinum neurotoxin type A were injected into the masseter muscles bilaterally (to a total of 50 units). A control group did not receive any intervention. MVBF was measured in Newtons using a strain gauge meter at the incisors and first molars. The intervention group was comprised of individuals seeking aesthetic treatment for masseter reduction (n = 20), and the control group (n = 12) comprised of volunteers.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects seeking aesthetical treatment to reduce masseter muscle volume.

Exclusion Criteria:

Conditions or drugs affecting the central nervous system.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Change of bite force | Baseline, 4 weeks, 3 months, 6 months, 12 months.
  Maximum voluntary bite force measured in Newtons at baseline, and change of bite force compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: 2020-03517 Pettersson, PhD, Principal Investigator — Umeå University
Locations (1):
- Norrlands universitetssjukhus, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No